CLINICAL TRIAL: NCT05771740
Title: Feasibility Study for Gathering Lung Sound Recordings From Pulmonary Fibrosis Patients and Healthy Controls and Classifying Disease Status Using a Combination of Digital Sound Device and Machine Learning
Brief Title: Pulmonary Fibrosis Lung Sounds Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2304409
Record Dates: First submitted 2023-01-30; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Fibrosis; Healthy
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary Fibrosis Patient: Participants under the clinical care of the interstitial lung disease team at the Royal Devon University Healthcare NHS Trust, UK
  Interventions: Device: Stemoscope (bluetooth sound amplifier)
- Healthy Control: Healthy participants visiting the Royal Devon University Healthcare NHS Trust, UK
  Interventions: Device: Stemoscope (bluetooth sound amplifier)

INTERVENTIONS:
Device: Stemoscope (bluetooth sound amplifier) — The bluetooth device will be placed in six locations on the front and six locations on the back of the chest and sound recordings stored for each location.

SUMMARY:
The goal of this observational study is to test whether it is possible to detect particular lung sounds that are unique to patients with the lung disease pulmonary fibrosis and whether any such sounds could be analysed using machine learning to make diagnosing disease easier.

Participants will have a sound detection device placed in different locations on the chest and audio sounds will be recorded for analysis.

Researchers will compare audio recordings from clinically diagnosed patients with recordings from healthy controls of a similar age to see whether the sounds are sufficiently different within that age group.

DETAILED DESCRIPTION:
This is a study of chest audio recordings obtained using a sound enhancer, in this case a Bluetooth device, combined with intelligent computer-processing and analysis. It is being carried out amongst pulmonary fibrosis patients and healthy controls of a similar age, with the aim to improve diagnosis of pulmonary fibrosis and remote monitoring of disease progression.

Expert respiratory doctors gain important insights about the health of a patient's lungs by listening to the chest with a stethoscope. Currently, there are insufficient respiratory experts and specialist equipment to meet the patient demand, leading to delays in diagnosis and treatment and a shortage of specialist care following diagnosis.

In this study the investigators are aiming to make that specialist practice much more available by recording lung sounds and developing software to do the intelligent analysis. Initial tests with publicly available recordings of expertly diagnosed respiratory sounds have shown that different lung diseases can be detected with a very high degree of accuracy using new software. Here the investigators want to test that software with a cost-effective digital sound device in a clinical setting. The aim is for respiratory diseases to be diagnosed quickly and easily and also, in future, for patients to be offered the option to monitor how well they are after diagnosis in their own home.

ELIGIBILITY:
Inclusion Criteria

* Able to understand what the study involves
* Able and willing to give informed consent

For patients:

* Age≥60 (PF affects adults, with the majority of age≥60)
* A diagnosis of progressive pulmonary fibrosis (to include all diagnosed interstitial lung disease (ILD) patients presenting at the ILD clinic)

For healthy controls:

* Age≥60 (to ensure that age of controls is similar to that of patients so that younger age does not bias results)
* No known lung disease

Exclusion Criteria

* Unable to understand what the study involves
* Unwilling or unable to give consent
* Age<60 (to ensure that age does not confound results and cases and controls are of similar age, since the majority of pulmonary fibrosis patients are of age≥60)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 50 Patients with a diagnosis of progressive pulmonary fibrosis attending routine interstitial lung disease clinic (age≥60) 50 Healthy controls of a similar age range (age≥60)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of clinical lung sound recordings stored from pulmonary fibrosis cases and controls | 6 months
  A measure of the feasibility of gathering 12 lung sound files from each of 50 PF patients and 50 healthy volunteers in a similar age-group in the available timeframe.
Measure of ability of this system to classify participants as PF patients or healthy controls | 8 months
  A measure of the capability of the machine learning model combined with the cost-effective bluetooth stethoscope to classify study participants as PF patients or healthy controls from lung sound recordings alone in a clinical setting
Feedback from patients and study clinicians | 8 months
  Feedback from patients and study clinicians about the acceptability of digital sound monitoring for improving future diagnosis and monitoring of disease progression in pulmonary fibrosis

SECONDARY OUTCOMES:
A correlation between clinical measures of pulmonary fibrosis severity and the audio waveform | 6 months
  A demonstrable correlation between objective markers of pulmonary function tests (forced vital capacity percent of predicted (FVC%) or diffusing capacity in the lung for carbon monoxide percentage predicted (DLCO%)) or breathlessness symptoms (mMRC Dyspnoea score) and the waveform of the audio recording.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gibbons, Principal Investigator — Royal Devon University Healthcare NHS Trust

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available on an anonymised basis via Open Research Exeter data depository (https://ore.exeter.ac.uk/repository).
Supporting Information: Study Protocol, ICF
Time Frame: In accordance with MRC data sharing policy, the anonymous electronic data will be stored indefinitely and will be available for sharing for research purposes on request after 2 years from receipt of the full dataset.
Access Criteria: Available on request as above
URL: http://ore.exeter.ac.uk/repository